CLINICAL TRIAL: NCT03108794
Title: A Nation-wide Hospital-based Hepatitis B Registry:China Registry of Hepatitis B
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Friendship Hospital (Other)
Collaborators: Beijing YouAn Hospital (Other); The First Hospital of Jilin University (Other); Henan Provincial People's Hospital (Other); Beijing Ditan Hospital (Other); First Affiliated Hospital of Xinjiang Medical University (Other); LanZhou University (Other); The Second Affiliated Hospital of Chongqing Medical University (Other); West China Hospital (Other); The Third People's Hospital of Taiyuan (Other); Hebei Medical University Third Hospital (Other); Shengjing Hospital (Other); Tianjin Third Central Hospital (Other); Peking University First Hospital (Other); Peking Union Medical College Hospital (Other); The Affiliated Hospital Of Southwest Medical University (Other); Shanghai Public Health Clinical Center (Other Government); Ruijin Hospital (Other); First Affiliated Hospital Xi'an Jiaotong University (Other); Xiangya Hospital of Central South University (Other); Beijing Tiantan Hospital (Other); Wuhan University (Other); First Affiliated Hospital of Kunming Medical University (Other); The Affiliated Hospital of Xuzhou Medical University (Other); The Affiliated Hospital of Yanbian University (Other); First Affiliated Hospital of Chongqing Medical University (Other); The Fourth People's Hospital of Qinghai Province (Other); Weifang Medical University (Other); Hunan Provincial People's Hospital (Other); The Second Hospital of Hebei Medical University (Other); Xixi Hospital of Hangzhou (Unknown); General Hospital of Ningxia Medical University (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Xinjiang Uygur Autonomous Region Traditional Chinese Medicine Hospital (Unknown); Peking University People's Hospital (Other); Nanfang Hospital, Southern Medical University (Other); The Affiliated Hospital Of Guizhou Medical University (Other); Guizhou Provincial People's Hospital (Other); Hainan General Hospital (Other); The Second Hospital of Shandong University (Other); The First Affiliated Hospital of Shanxi Medical University (Other); Fifth Hospital of Shijiazhuang City (Other); Yan'an University Affiliated Hospital (Other); Infectious Disease Hospital of Wuhai (Unknown); Logistics University of Chinese People's Armed Police Forces (Other); People's Hospital of Changji Hui Autonomous Prefecture，Xinjiang (Unknown)
Responsible Party: Principal Investigator, Jidong Jia, Liver Research Center, Beijing Friendship Hospital
Other Study IDs: CR-HepB
Record Dates: First submitted 2017-04-06; First posted 2017-04-11 (Actual); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Chronic Hepatitis B
Keywords: hepatitis B，registry,cirrhosis, HCC
MeSH Terms: conditions — Hepatitis B, Chronic; Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- Immune tolerance phase: Immune tolerance phase is diagnosed based on the presence of high serum levels of HBV-DNA, hepatitis B e antigen (HBeAg), but normal or minimally elevated serum alanine aminotransferase (ALT), and normal liver or only minimal histological activity and scant fibrosis.
- HBeAg positive CHB: HBeAg positive CHB is defined as those with HBsAg positive for more 6 months, HBeAg positive, high HBV DNA, elevated serum levels of ALT and histological activity.
- HBeAg negative CHB: HBeAg negative CHB is defined as those with HBeAg negative, anti-HBe positive, lower serum HBV DNA levels and histological necroinflammation and fibrosis.
- Inactive HBsAg carriers: Inactive HBsAg carriers was defined as those with HBsAg positive than 6 months, with low HBV DNA and persistently normal ALT, without evidence of cirrhosis.
- Compensated cirrhosis: Diagnosis of compensated cirrhosis can be made if one of the following criteria was met:
  1. by liver histology: Ishak fibrosis stage 5-6 or METAVIR F4.
  2. endoscopy-proven gastroesophageal varices, afrter excluding non-cirrhotic portal hypertension.
  3. at least 2 features of cirrhosis:
     1. irregular liver surface, granular or nodular liver parenchyma, with or without splenomegaly (spleen thickness > 4.0cm or > 5 rib units) on ultrasound ,CT or MRI;
     2. PLT<100×109/L without other causes;
     3. Serum album in<35 g/L or INR>1.3 or PT prolongs>3s;
     4. LSM>13 kpa (ALT<5×ULN).
- Decompensated cirrhosis: Decompensated cirrhosis was diagnosed based on the presence of ascites, bleeding esophageal varices and/or hepatic encephalopathy in cirrhotic patients.
- Hepatocellular carcinoma: Diagnosis of hepatocellular carcinoma（HCC）can be established when one of the following one of the following 2 criteria:（1）in cirrhotic patients with nodules of 1cm or larger with typical features of HCC ( arterial enhancement with washout in venous or delay phase) on 2 radiological studies or with 1 radiological study and elevation of serum AFP; or（2）histological evidence of HCC.

SUMMARY:
CR-HepB registry started in June 30,2012 to collect HBV cases from general hospitals or specialized hospitals for infectious diseases in mainland China. Demographics, diagnosis, laboratory test results, family history and prescriptions were recorded. The main criteria for registration is HBsAg-positivity more than 6 months, and these patients will receive followed-up visits every three to six months.

DETAILED DESCRIPTION:
This web-based database was launched on June 30, 2012 and consists of tertiary or secondary hospitals with special interest and expertise on managing hepatitis B patients across mainland China. The main inclusion criteria for this registration are HBsAg-positivity ≥ 6 months, HBeAg positive or negative, with or without cirrhosis, either treatment-naïve or treatment experienced. At the first time of data entry, demographics, medical history, virology, biochemistry and hematology results, radiology reports, diagnosis and treatment information were recorded. Then the registered patients received standard of care and follow-up every 3 to 6 months. On each visit, virological, biochemical, and radiological reports, as well as clinical progress were recorded.

ELIGIBILITY:
Inclusion Criteria:

* HBsAg-positivity over a continuous six months.

The core exclusion criteria are: 1) HCC patients for their treatment mainly depends on surgical operation and interventional therapy, but not the antiviral therapy; 2) patients who are unable or unwilling to provide informed consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The registry is a multicentre and observational study enrolling patients with hepatitis B across China. The main criteria for patients registration within the system was HBsAg-positivity over a continuous six months. The core exclusion criteria are: 1) HCC patients for their treatment mainly depends on surgical operation and interventional therapy, but not the antiviral therapy; 2) patients who are unable or unwilling to provide informed consent. All potential subjects meeting enrollment criteria are offered the opportunity to participate.
Sampling Method: Non-Probability Sample
Enrollment: 200000 (Estimated)
Dates: Start 2012-06-30 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of liver-related events after antiviral therapy | 10 years
  Rates of cirrhosis,decompensation and hepatocellular carcinoma with or without antiviral therapy

SECONDARY OUTCOMES:
The HBV DNA undetectable rate with or without antiviral therapy | 10 years
HBeAg loss and seroconversion rates with or without antiviral therapy | 10 years

OTHER OUTCOMES:
HBsAg loss and seroconversion rates with or without antiviral therapy | 10 years
Quality of life | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Jidong Jia, Doctor, Principal Investigator — Beijing Friendship Hospital
Locations (45):
- China (45):
  - Beijing Ditan Hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Beijing Tiantan Hospital, Beijing, Beijing Municipality
  - Beijing Youan Hospital, Beijing, Beijing Municipality
  - The Second Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Lanzhou University Second Hospital, Lanzhou, Gansu
  - The First Hospital of Lanzhou University, Lanzhou, Gansu
  - Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong
  - The Affiliated Hospital of Guizhou Medical University, Guiyang, Guizhou
  - Guizhou provincial people's hospital, Guiyang, Guizhou
  - Hainan General Hospital, Haikou, Hainan
  - The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The Fifth Hospital of Shijiazhuang, Shijiazhuang, Hebei
  - The Third Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - Union Hospital,Tong Ji Medical College,Huazhong University of Science and Technology, Wuhan, Hubei
  - Zhongnan Hospital of Wuhan University, Wuhan, Hubei
  - Hunan Provincial People's Hospital, Changsha, Hunan
  - Xiangya Hospital Central South University, Changsha, Hunan
  - Infectious Disease Hospital of Wuhai, Wuhai, Inner Mongolia
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - First Hospital of Jilin University, Changchun, Jilin
  - The Affiliated Hospital of Yanbian University, Yanbian, Jilin
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - General Hospital of Ningxia Medical University, Yinchuan, Ningxia
  - The Second Hospital of Shandong University, Jinan, Shandong
  - Affiliated Hospital of Weifang Medical University, Weifang, Shandong
  - Shanghai Ruijin Hospital, Shanghai, Shanghai Municipality
  - Shanghai Public Health Clinical Center, Shanghai, Shanghai Municipality
  - The First Affiliated Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Taiyuan No.3 Hospital, Taiyuan, Shanxi
  - First Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi
  - Yanan University Affiliated Hospital, Yanan, Shanxi
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - The Affiliated Hospital of Southwest Medical University, Luzhou, Sichuan
  - Affiliated Hospital, Logistics University of People's Armed Police Force, Tianjin, Tianjin Municipality
  - Tianjin Third Central Hospital, Tianjin, Tianjin Municipality
  - People's Hospital of Changji Hui Autonomous Prefecture，Xinjiang, Changji, Xinjiang
  - First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - Xinjiang Uygur Autonomous Region Traditional Chinese Medicine Hospital, Ürümqi, Xinjiang
  - First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - Xixi Hospital of Hangzhou, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] You H, Kong Y, Hou J, Wei L, Zhang Y, Niu J, Han T, Ou X, Dou X, Shang J, Tang H, Xie Q, Ding H, Ren H, Xu X, Xie W, Liu X, Xu Y, Li Y, Li J, Chow SC, Zhuang H, Jia J. Female gender lost protective effect against disease progression in elderly patients with chronic hepatitis B. Sci Rep. 2016 Nov 28;6:37498. doi: 10.1038/srep37498. PMID 27892487
- [Derived] Zhang Y, Wang Y, Jiao S, Li S, Liu X, Li T, Qu Y. Nonlinear relationship between age and the risk of hepatocellular carcinoma in patients with hepatitis B virus-related cirrhosis. BMC Infect Dis. 2025 Nov 21;25(1):1635. doi: 10.1186/s12879-025-12016-9. PMID 41272517
- [Derived] Shan S, Wei W, Kong Y, Niu J, Shang J, Xie W, Zhang Y, Ren H, Tang H, Ding H, Nan Y, Dou X, Han T, Xu X, Duan Z, Wei L, Hou J, Zhuang H, You H, Jia J; CR-Hepb Study Group, Beijing, China. China Registry of Hepatitis B (CR-HepB): Protocol and implementation of a nationwide hospital-based registry of hepatitis B. Scand J Public Health. 2020 Mar;48(2):233-239. doi: 10.1177/1403494818772188. Epub 2018 May 1. PMID 29716439